CLINICAL TRIAL: NCT03830099
Title: Inhomogeneous Ventilation in Adult Post-neurosurgical Patients: an Observational Study
Brief Title: Inhomogeneous Ventilation in Adult Post-neurosurgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Other Study IDs: KY 2018-006-01
Record Dates: First submitted 2019-01-29; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Mechanical Ventilation; Electrical Impedance Tomography; Inhomogeneous Ventilation; Neurosurgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inhomogeneous ventilation was more likely to happen in patients after general anesthesia. Inhomogeneous ventilation may associate with ventilator-induced lung injury. A large number of post-neurosurgical patients was delayed extubation and received mechanical ventilation, so that, inhomogeneous ventilation was more likely to happen in the population. Electrical impedance tomography (EIT) is an noninvasive, radiation-free, high temporal resolution, relatively cheap technique in monitoring ventilation distribution bedside. The investigators aimed to investigate the incidence of inhomogeneous ventilation and factors associated with inhomogeneous ventilation in post-neurosurgical patients under mechanical ventilation.

DETAILED DESCRIPTION:
Inhomogeneous ventilation was more likely to happen in patients after general anesthesia. Inhomogeneous ventilation may associate with ventilator-induced lung injury since the gravity-depend collapse and over-distention of nondependent regional in patients under mechanical ventilation. A large number of post-neurosurgical patients was delayed extubation and received mechanical ventilation, so that, inhomogeneous ventilation was more likely to happen in the population. Up to now, there is no research reported about the prevalence of inhomogeneous ventilation and the factors associated with inhomogeneous ventilation in post-neurosurgical patients, in present study, The investigators prospectively enrolled adult patients after neurosurgical operations. Electrical impedance tomography (EIT) is an noninvasive, radiation-free, high temporal resolution, relatively cheap technique in monitoring ventilation distribution bedside. The investigators aimed to investigate the incidence of inhomogeneous ventilation and factors associated with inhomogeneous ventilation in post-neurosurgical patients under mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective neurosurgery operation
* Trachea intubated and mechanical ventilated

Exclusion Criteria:

* Age under 18 years-old
* Unstable hemodynamics patients (mean arterial pressure under 65mmHg) after pharmacotherapy
* History of chronic obstructive pulmonary disease(COPD) or asthma
* Contraindication of using EIT (pacemaker, defibrillator, and implantable pumps)
* Unable to install EIT belt (skin infection, wound)
* Incompleteness of thorax (e.g. pneumothorax, rib fracture and etc.) or malformation of thorax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender was based on basic information collected at the moment when patients was admitted to hospital.
Study Population: Adult post-neurosurgical patients under mechanical ventilation(MV).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of inhomogeneous ventilation | within 24 hours after neurosurgical operative
  In supine position, global image of EIT was divided into upper and lower part, each part accounting for 50%, which was named as non-dependent region and dependent region respectively. Inhomogeneous ventilation was defined as the ratio between tidal impedance variation of dependent region(VTdep) and global tidal impedance variation (VT) is less than 45% during stable Spontaneous breath, which was defined as variation of tidal volume less than 10% in continuous 6 breathes.

SECONDARY OUTCOMES:
The incidence of postoperative pulmonary complications(PPCs) | 28 days after neurosurgical operative
  Postoperative pulmonary complication was defined as follows: Pneumonia was defined as recent pulmonary infiltration on chest radiography associated with at least 2 of the following signs: purulent tracheobronchial secretion, a body temperature > 38.3℃，and leukocytes in peripheral blood > 25% above the basal count. Tracheobronchitis was an increase in the volume or a change in the color or purulent aspect of tracheobronchial secretion with a normal chest radiograph. Atelectasis was evidence on chest radiography of pulmonary atelectasis associated with acute respiratory symptoms. Bronchoconstriction was classified as the presence of wheezing associated with acute respiratory symptoms with a good response to inhalatory bronchodilator medication.
Length of ICU stay | through study completion, an average of 7 days
  The number of days that patients stay in ICU.
Length of hospital stay | through study completion, an average of 28 days
  The number of days that patients stay in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China